CLINICAL TRIAL: NCT03259373
Title: IMplementation of a Randomized Controlled Trial (RCT) to imProve Treatment With Oral AntiCoagulanTs in Patients With Atrial Fibrillation
Brief Title: IMplementation of an RCT to imProve Treatment With Oral AntiCoagulanTs in Patients With Atrial Fibrillation
Acronym: IMPACT-AFib
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Duke Clinical Research Institute (Other); Clinical Trials Transformation Initiative (Other); Humana Inc. (Industry); Aetna, Inc. (Industry); OptumInsight Life Sciences, Inc. (Unknown); Food and Drug Administration (FDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Richard Platt, Professor and Department Chair, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IMPACT-AFib
Record Dates: First submitted 2017-07-07; First posted 2017-08-23 (Actual); Results first posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Atrial Fibrillation; Stroke
Keywords: AF; AFib; OAC; Atrial fibrillation; Oral anticoagulant; Education
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Educational mailing to (1) AF patients with guideline-based indications for oral anticoagulation (CHA₂DS₂-VASc score of 2 or greater) who appear to not have received OAC treatment at time of randomization and (2) their providers, where an individual provider may be identified
  Interventions: Behavioral: Early Patient-Level and Provider-Level Educational Intervention
- Control (Experimental): Educational mailing to providers of AF patients with guideline-based indications for oral anticoagulation (CHA₂DS₂-VASc score of 2 or greater) who appear to not have received OAC treatment in the time following randomization. These patients will have received 'usual care' for the time between randomization and delayed educational mailing.
  Interventions: Behavioral: Delayed Provider-Level Educational Intervention

INTERVENTIONS:
Behavioral: Early Patient-Level and Provider-Level Educational Intervention — Letters to patients that (1) explain to the patient that he or she appears to have AF, characterize the risk of stroke, and emphasize that although there may be a medical reason, the patient does not seem to be on an anticoagulant and (2) encourage the patient to discuss this with his or her provider to ask if he or she might benefit from OAC therapy to prevent stroke.
  Early intervention letters to providers explain this project, the nature of the problem, and identify a list of the provider's patients who have been contacted, as the provider and patient letters will be sent at approximately the same time; describe evidence and guidelines regarding oral anticoagulation.
  Arms: Intervention
Behavioral: Delayed Provider-Level Educational Intervention — Delayed intervention letters to patients' providers, where they may be identified, that explain this project, the nature of the problem, and identify a list of their patients who are flagged as at risk for stroke and have not been treated with an oral anticoagulant; describe evidence and guidelines regarding oral anticoagulation.
  Arms: Control

SUMMARY:
The purpose of this study is to use a decentralized claims database to determine whether education on stroke prevention in atrial fibrillation (AF) among AF patients and their providers can result in increased use of oral anticoagulants (OAC) for stroke prevention among those AF patients with guideline-based indications for oral anticoagulation (CHA₂DS₂-VASc score of 2 or greater). Specifically, the investigators will conduct a prospective, randomized, open-label education intervention trial to evaluate the effect of the early patient and provider education interventions on the proportion of patients with evidence of at least one OAC prescription fill (defined as one OAC dispensing or 4 international normalized ratio [INR tests] over the course of the follow-up through the date on which at least 80% of eligible study participants have at least 12 months of follow-up time). A total of approximately 80,000 patients will be enrolled within multiple major health plans across the United States. The randomization will be performed by the central coordinating center, and the health plans will mail the educational intervention materials to their members and providers.

DETAILED DESCRIPTION:
The study is a prospective, randomized, and open-label education intervention trial. Patients with AF and a CHA₂DS₂-VASc score of 2 or greater will be randomized in a 1:1 ratio to an intervention cohort and a control cohort within each participating health plan. The definition for OAC medication fill will be an OAC medication dispensing or at least 4 INR tests in the claims data. The claims records of the patients randomized to the intervention cohort will then be linked to "fresh" (i.e. about 1 month old) pharmacy claims data at the time of randomization. Patients without evidence of an OAC medication fill during the 12 months prior to randomization will be included in the patient-level and provider-level early educational intervention. In addition to usual care, these patients and their providers, where an individual provider may be identified, will receive a one-time mailing at trial start. Patients randomized to this early intervention with evidence of an OAC medication fill during the 12 months prior to randomization will be excluded from the trial.

The control cohort will receive usual care over the initial study period. After the date on which at least 80% of eligible study participants have at least 12 months of follow-up time, "fresh" pharmacy claims data for the control intervention cohort that was generated and locked at the time of randomization will be used to assess trial eligibility, and those patients without evidence of an OAC medication fill during the 12 months prior to randomization will be included in the primary and secondary analyses as the control arm. Patients randomized to the control arm with evidence of an OAC medication fill during the 12 months prior to randomization will be excluded from the trial and will not be included in analyses. The baseline characteristics of the control patients will be examined at the same time point as the intervention patients, meaning at the time of randomization. The primary outcome is a comparison of the proportion of patients not on OAC during the 12 months prior to randomization, who were started on OAC over the course of the follow-up through the date on which at least 80% of eligible study participants have at least 12 months of follow-up time in the early versus the delayed intervention arm. A total of approximately 80,000 patients (randomized 1:1) across all participating data partners (Aetna, Harvard Pilgrim, Humana, and Optum) will be enrolled from participating data partners across the United States. The follow-up time for the primary outcome will be 12 months from the date at which at least 80% of eligible study participates are enrolled (date on which early intervention materials are mailed).

The providers of patients in the control cohort who did not receive OAC medication during the course of the 12-month study period and meet the inclusion criteria will receive the delayed intervention: the provider-only education intervention, a one-time mailing administered 12 months after at least 80% of early intervention mailings have occurred (patients will not receive any educational materials). The investigators intend to assess the primary and secondary endpoints again 24 months after at least 80% of early intervention mailings have occurred to assess the durability and longer-term outcomes of the effect of the patient- and provider-level education intervention, as well as the use of OAC following the delayed provider-level education intervention. However, as this second assessment is exploratory, investigators may not conduct these analyses if the results of the primary outcome are consistently null.

Because the Sentinel Distributed Database will be used for follow-up information, and this information is refreshed approximately quarterly and this is done on separate timetables for the different health plans, it is likely that when at least the required follow-up time is available for at least 80% of people, there will be more than 12 or 24 months of followup for over 80% of people. All participants' outcomes will be assessed using all possible person-time; patients will have different duration of follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Two or more diagnoses of AF (ICD-9 and/or 10 codes) at least one day apart and with at least one diagnosis within the last 12 months prior to the last date in the current approved data used for cohort identification
2. CHA₂DS₂-VASc score of 2 or greater
3. Medical and pharmacy insurance coverage of at least the prior year as identified via administrative claims databases of one of the participating data partners as of the date of randomization
4. Age 30 years or greater as of the last date in the current approved data used for cohort identification

Exclusion Criteria:

1. Evidence of OAC medication fill during the 12 months prior to randomization (determined at randomization for the early intervention cohort and 12 months post-randomization for the delayed intervention cohort)
2. Conditions other than AF that require anticoagulation, including treatment of deep venous thrombosis, pulmonary embolism, or ever having had a mechanical prosthetic heart valve prior to the last date in the current approved data used for cohort identification
3. Pregnancy within 6 months of the last date in the current approved data used for cohort identification
4. Any known history of intracranial hemorrhage prior to the last date in the current approved data used for cohort identification
5. Hospitalization for bleeding within the last 6 months of the last date in the current approved data used for cohort identification
6. Patients with recent P2Y12 antagonist use (i.e. clopidogrel, prasugrel, ticlopidine, or ticagrelor within 90 days of the last date in the current approved data used for cohort identification

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64666 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Humana Healthcare Research, Inc., Louisville, Kentucky
  - Harvard Pilgrim Health Care, Quincy, Massachusetts
  - OptumInsight, Inc, Waltham, Massachusetts
  - Aetna, Inc., Blue Bell, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pokorney SD, Cocoros N, Al-Khalidi HR, Haynes K, Li S, Al-Khatib SM, Corrigan-Curay J, Driscoll MR, Garcia C, Calvert SB, Harkins T, Jin R, Knecht D, Levenson M, Lin ND, Martin D, McCall D, McMahill-Walraven C, Nair V, Parlett L, Petrone A, Temple R, Zhang R, Zhou Y, Platt R, Granger CB. Effect of Mailing Educational Material to Patients With Atrial Fibrillation and Their Clinicians on Use of Oral Anticoagulants: A Randomized Clinical Trial. JAMA Netw Open. 2022 May 2;5(5):e2214321. doi: 10.1001/jamanetworkopen.2022.14321. PMID 35639381
- [Derived] Garcia CJ, Haynes K, Pokorney SD, Lin ND, McMahill-Walraven C, Nair V, Parlett L, Martin D, Al-Khalidi HR, McCall D, Granger CB, Platt R, Cocoros NM. Practical challenges in the conduct of pragmatic trials embedded in health plans: Lessons of IMPACT-AFib, an FDA-Catalyst trial. Clin Trials. 2020 Aug;17(4):360-367. doi: 10.1177/1740774520928426. Epub 2020 Jun 26. PMID 32589056
- See also: White Paper: Developing Approaches to Conducting Randomized Trials Using the Mini-Sentinel Distributed Database — https://www.sentinelinitiative.org/sites/default/files/Methods/Mini-Sentinel_Methods_CTTI_Developing-Approaches-to-Conducting-Randomized-Trials-Usi.pdf
- See also: Sentinel Initiative IMPACT-AFib Project Page — https://www.sentinelinitiative.org/FDA-catalyst/projects/implementation-randomized-controlled-trial-improve-treatment-oral-anticoagulants-patients

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients and their treating clinicians were identified through health insurance claims data from commercially-insured and Medicare Advantage populations.
Groups:
- Intervention: Educational mailing to (1) AF patients with guideline-based indications for oral anticoagulation (CHA₂DS₂-VASc score of 2 or greater) who appear to not have received OAC treatment at time of randomization and (2) their providers, where an individual provider may be identified
  Early Patient-Level and Provider-Level Educational Intervention: Letters to patients that (1) explain to the patient that he or she appears to have AF, characterize the risk of stroke, and emphasize that although there may be a medical reason, the patient does not seem to be on an anticoagulant and (2) encourage the patient to discuss this with his or her provider to ask if he or she might benefit from OAC therapy to prevent stroke.
  Early intervention letters to providers explain this project, the nature of the problem, and identify a list of the provider's patients who have been contacted, as the provider and patient letters will be sent at approximately the same time; describe evidence and guidelines regarding oral anticoagulation.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 32295 | 32371
Completed | 23546 | 23787
Not Completed | 8749 | 8584
Not completed — Evidence of OAC treatment prior to start date based on more complete data | 636 | 118
Not completed — Disenrolled earlier than originally captured in data (due to changing in data over time) | 320 | 344
Not completed — Unable to be identified in dataset used for analysis | 43 | 49
Not completed — Censored between old dataset and the follow-up start date (due to changing in data over time) | 3446 | 3599
Not completed — Censored prior to old dataset, other reason (unable to specify reason from available data) | 32 | 63
Not completed — On OAC treatment at follow up start (due to data lags) | 4272 | 4411

BASELINE CHARACTERISTICS:
Groups:
- Intervention: Educational mailing to (1) AF patients with guideline-based indications for oral anticoagulation (CHA₂DS₂-VASc score of 2 or greater) who appear to not have received OAC treatment at time of randomization and (2) their providers, where an individual provider may be identified.
  Early Patient-Level and Provider-Level Educational Intervention: Letters to patients that (1) explain to the patient that he or she appears to have AF, characterize the risk of stroke, and emphasize that although there may be a medical reason, the patient does not seem to be on an anticoagulant and (2) encourage the patient to discuss this with his or her provider to ask if he or she might benefit from OAC therapy to prevent stroke.
  Early intervention letters to providers explain this project, the nature of the problem, and identify a list of the provider's patients who have been contacted, as the provider and patient letters will be sent at approximately the same time; describe evidence and guidelines regarding oral anticoagulation.
- Control: Delayed Provider-Level Educational Intervention: The control arm patients received "usual care" for the time between randomization and a delayed educational mailing, which was sent after one year.
  Delayed intervention included the following:
  Educational mailing to providers of AF patients with guideline-based indications for oral anticoagulation (CHA₂DS₂-VASc score of 2 or greater) who appear to not have received OAC treatment in the time following randomization. These letters to patients' providers, where they may be identified, explain this project, the nature of the problem, and identify a list of their patients who are flagged as at risk for stroke and have not been treated with an oral anticoagulant; describe evidence and guidelines regarding oral anticoagulation.
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 23,546 | 23,787 | 47333
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.8 (9.7) | 77.9 (9.7) | 77.8 (9.7)
Age, Customized [Count of Participants; unit: Participants]
  Age < 55 yr | 471 | 436 | 907
  Age 55-59 yr | 569 | 562 | 1131
  Age 60-64 yr | 934 | 979 | 1913
  Age 65-69 yr | 2,341 | 2,360 | 4701
  Age 70-74 yr | 4,642 | 4,762 | 9404
  Age 75-79 yr | 4,814 | 4,946 | 9760
  Age 80-84 yr | 4,182 | 3,966 | 8148
  Age 85-89 yr | 3,169 | 3,205 | 6374
  Age 90 and older | 2,424 | 2,571 | 4995
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11,262 | 11,162 | 22424
  Male | 12,284 | 12,625 | 24909
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States: New England | 645 | 731 | 1376
  United States: Mid-Atlantic | 1,162 | 1,298 | 2460
  United States: South-Atlantic | 14,340 | 14,286 | 28626
  United States: Midwest | 4,723 | 4,885 | 9608
  United States: Mountain | 1,484 | 1,470 | 2954
  United States: Pacific | 906 | 859 | 1765
  United States: Unknown/missing | 286 | 258 | 544
History of hypertension [Count of Participants; unit: Participants] | 22,338 | 22,583 | 44921
History of diabetes [Count of Participants; unit: Participants] | 9,671 | 9,625 | 19296
History of peripheral vascular disease [Count of Participants; unit: Participants] | 6,001 | 5,981 | 11982
History of prior cerebrovascular disease [Count of Participants; unit: Participants] | 4,944 | 4,863 | 9807
History of heart failure [Count of Participants; unit: Participants] | 9,451 | 9,452 | 18903
History of MI [Count of Participants; unit: Participants] | 2,827 | 2,744 | 5571
History of CABG [Count of Participants; unit: Participants] | 3,409 | 3,500 | 6909
History of coronary stent [Count of Participants; unit: Participants] | 1,205 | 1,188 | 2393
Dialysis [Count of Participants; unit: Participants] | 664 | 616 | 1280
CHA2DS2-VASc score, mean [Mean (Standard Deviation); unit: units on a scale] — The CHA2DS2-VASc score, which ranges from 0 (minimum) to 9 (maximum), is a point-based system used to stratify the risk of stroke in atrial fibrillation (AF) patients. Patients with a score of 0 have low risk of stroke, patients with a score of 1 have intermediate risk of stroke, and patients with a score of 2 or more are at high risk of stroke.
  units on a scale | 4.53 (1.7) | 4.50 (1.7) | 4.51 (1.7)
ATRIA Score ≥ 5 [Count of Participants; unit: Participants] | 11,165 | 11,239 | 22404
History of hospitalization for bleeding [Count of Participants; unit: Participants] | 4,409 | 4,481 | 8890

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Evidence of at Least One OAC Dispensing (Prescription Fill) (Defined as One OAC Dispensing or 4 INR (International Normalized Ratio) Tests)
Description: Evaluate the effect of the patient and provider education interventions (versus usual care with delayed provider education intervention) on the proportion of patients with evidence of at least one OAC prescription fill (defined as one OAC dispensing or 4 INR tests) over the course of the 12 months of follow-up.
Time Frame: Outcome assessed at 42 days, 90 days, 183 days, and one year of follow-up time.
Population: Overall number of participants, as well as prespecified sex, age, and CHA2DS2-VASC score subgroups.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 23,546 | 23,787
Participants
  OAC initiation at one year (primary) | 2,328 | 2,330
  OAC initiation at 183 days | 1403 | 1362
  OAC initiation at 90 days | 769 | 738
  OAC initiation at 42 days | 394 | 361
  OAC initiation at one year, female: number analyzed (Participants) | 11,262 | 11,162
  OAC initiation at one year, female | 1,146 | 1,081
  OAC initiation at one year, male: number analyzed (Participants) | 12,284 | 12,625
  OAC initiation at one year, male | 1,182 | 1,249
  OAC initiation at one year, age <65 years: number analyzed (Participants) | 1,443 | 1,474
  OAC initiation at one year, age <65 years | 141 | 145
  OAC initiation at one year, age 65-74 years: number analyzed (Participants) | 6,755 | 6,911
  OAC initiation at one year, age 65-74 years | 704 | 707
  OAC initiation at one year, age 75-84 years: number analyzed (Participants) | 8,927 | 8,823
  OAC initiation at one year, age 75-84 years | 987 | 954
  OAC initiation at one year, age >=85: number analyzed (Participants) | 5,560 | 5,740
  OAC initiation at one year, age >=85 | 424 | 440
  OAC initiation at one year, CHA2DS2-VASC score of 2-3: number analyzed (Participants) | 7,073 | 7,183
  OAC initiation at one year, CHA2DS2-VASC score of 2-3 | 657 | 683
  OAC initiation at one year, CHA2DS2-VASC score of 4-5: number analyzed (Participants) | 10,150 | 10,397
  OAC initiation at one year, CHA2DS2-VASC score of 4-5 | 1,041 | 992
  OAC initiation at one year, CHA2DS2-VASC score >=6: number analyzed (Participants) | 6,309 | 6,183
  OAC initiation at one year, CHA2DS2-VASC score >=6 | 629 | 654
Statistical Analysis 1: Comparison: Intervention vs Control; The null hypothesis was the that proportions of patients with at least one OAC filled at one year were the same between the two groups; Test type: Superiority; p = 0.79, fixed-effect meta-analysis; Odds Ratio (OR) = 1.01, 95% CI 2-sided [0.95 to 1.07], Standard Error of Mean 0.031
Statistical Analysis 2: Comparison: Intervention vs Control; The null hypothesis was that the proportions of patients with at least one OAC filled at 183 days were the same between the two groups; Test type: Superiority; p = 0.307, fixed-effect meta-analysis; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.96 to 1.12], Standard Error of Mean 0.039
Statistical Analysis 3: Comparison: Intervention vs Control; The null hypothesis was that the proportions of patients with at least one OAC filled at 90 days were the same between the two groups; Test type: Superiority; p = 0.375, fixed-effect meta-analysis; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.95 to 1.16], Standard Error of Mean 0.052
Statistical Analysis 4: Comparison: Intervention vs Control; The null hypothesis was that the proportions of patients with at least one OAC filled at 42 days were the same between the two groups; Test type: Superiority; p = 0.265, fixed-effect meta-analysis; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.94 to 1.26], Standard Error of Mean 0.076
Statistical Analysis 5: Comparison: Intervention vs Control; The null hypothesis was that the proportions of patients with at least one OAC filled among females were the same between the two groups; Test type: Superiority; p = 0.237, fixed-effect meta-analysis; Odds Ratio (OR) = 1.05, 95% CI 2-sided [0.97 to 1.15], Standard Error of Mean 0.044
Statistical Analysis 6: Comparison: Intervention vs Control; The null hypothesis was that the proportions of patients with at least one OAC filled among males were the same between the two groups; Test type: Superiority; p = 0.487, fixed-effect meta-analysis; Odds Ratio (OR) = 0.97, 95% CI 2-sided [0.89 to 1.05], Standard Error of Mean 0.042
Statistical Analysis 7: Comparison: Intervention vs Control; The null hypothesis was that the proportions of patients with at least one OAC filled among age <= 64 yrs were the same between the two groups; Test type: Superiority; p = 0.952, fixed-effect meta-analysis; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.78 to 1.27], Standard Error of Mean 0.125
Statistical Analysis 8: Comparison: Intervention vs Control; The null hypothesis was that the proportions of the patients with at least one OAC filled among age 65 - 74 yrs were the same between the two groups; Test type: Superiority; p = 0.696, fixed-effect meta-analysis; Odds Ratio (OR) = 1.02, 95% CI 2-sided [0.91 to 1.14], Standard Error of Mean 0.057
Statistical Analysis 9: Comparison: Intervention vs Control; The null hypothesis was that the proportions of patients with at least one OAC filled among age 75 - 84 yrs were the same between groups; Test type: Superiority; p = 0.584, fixed-effect meta-analysis; Odds Ratio (OR) = 1.03, 95% CI 2-sided [0.94 to 1.13], Standard Error of Mean 0.047
Statistical Analysis 10: Comparison: Intervention vs Control; The null hypothesis was that the proportions of patients with at least one OAC filled among age >= 85 yrs were the same between the two groups; Test type: Superiority; p = 0.911, fixed-effect meta-analysis; Odds Ratio (OR) = 0.99, 95% CI 2-sided [0.87 to 1.14], Standard Error of Mean 0.069
Statistical Analysis 11: Comparison: Intervention vs Control; The null hypothesis was that the proportions of the patients with at least one OAC filled among those with a CHADS-VASC of 2-3 were the same between the two groups; Test type: Superiority; p = 0.746, fixed-effect meta-analysis; Odds Ratio (OR) = 0.98, 95% CI 2-sided [0.88 to 1.10], Standard Error of Mean 0.057
Statistical Analysis 12: Comparison: Intervention vs Control; The null hypothesis was that the proportions of patients with at least one OAC filled among those with a CHADS-VASC score of 4-5 were the same between the two groups; Test type: Superiority; p = 0.109, fixed-effect meta-analysis; Odds Ratio (OR) = 1.08, 95% CI 2-sided [0.98 to 1.19], Standard Error of Mean 0.048
Statistical Analysis 13: Comparison: Intervention vs Control; The null hypothesis was that the proportions of patients with at least one OAC filled among those with a CHADS-VASC score >=6 were the same between the two groups; Test type: Superiority; p = 0.244, fixed-effect meta-analysis; Odds Ratio (OR) = 0.94, 95% CI 2-sided [0.84 to 1.05], Standard Error of Mean 0.057

2. Secondary Outcome: Rates of Hospitalization for Ischemic or Unknown Stroke
Description: Evaluate the impact of the patient and provider education interventions on rates of ischemic / unknown stroke hospitalization
Time Frame: Outcome assessed at one year of follow-up time.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 23,267 | 23,503
Participants | 341 | 375
Statistical Analysis 1: Comparison: Intervention vs Control; There were one or two sites that had no adverse events or just one event in either or both arms, so there was no estimated effect size/variance from the multivariable models at the site level. Therefore, depending on the specific outcome, either one or two sites did not contribute to the fixed-effect meta-analysis as there was no estimated effect size or variance to include in the meta-analysis; Test type: Superiority; p = 0.300, fixed-effect meta-analysis; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.79 to 1.08], Standard Error of Mean 0.079

3. Secondary Outcome: Rates of Hospitalization for Hemorrhagic Stroke
Description: Evaluate the impact of the patient and provider education interventions on rates of hospitalization for hemorrhagic stroke
Time Frame: Outcome assessed at one year of follow-up time.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 22,685 | 22,948
Participants | 81 | 64
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.122, fixed-effect meta-analysis; Hazard Ratio (HR) = 1.31, 95% CI 2-sided [0.93 to 1.83], Standard Error of Mean 0.172

4. Secondary Outcome: Rates of Hospitalization for Ischemic or Hemorrhagic Stroke
Description: Evaluate the impact of the patient and provider education interventions on rates of hospitalization for ischemic or hemorrhagic stroke
Time Frame: Outcome assessed at one year of follow-up time.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 23,267 | 23,503
Participants | 419 | 436
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.760, fixed-effect meta-analysis; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.85 to 1.13], Standard Error of Mean 0.073

5. Secondary Outcome: Rates of Hospitalization for Ischemic or Hemorrhagic Stroke or Systemic Embolism
Description: Evaluate the impact of the patient and provider education interventions on rates of hospitalization for ischemic or hemorrhagic stroke or systemic embolism
Time Frame: Outcome assessed at one year of follow-up time.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 23,267 | 23,503
Participants | 441 | 453
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.760, fixed-effect meta-analysis; Hazard Ratio (HR) = 0.99, 95% CI 2-sided [0.86 to 1.14], Standard Error of Mean 0.072

6. Secondary Outcome: Rates of Hospitalization for Ischemic or Hemorrhagic Stroke or Systemic Embolism or Bleeding
Description: Evaluate the impact of the patient and provider education interventions on rates of hospitalization for ischemic or hemorrhagic stroke or systemic embolism or bleeding
Time Frame: Outcome assessed at one year of follow-up time.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 23,267 | 23,503
Participants | 733 | 760
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.616, fixed-effect meta-analysis; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.88 to 1.08], Standard Error of Mean 0.052

7. Secondary Outcome: Rates of Hospitalization for Bleeding
Description: Evaluate the impact of the patient and provider education interventions on rates of hospitalization for any bleeding
Time Frame: Outcome assessed at one year of follow-up time.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 22,685 | 22,948
Participants | 382 | 385
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.992, fixed-effect meta-analysis; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.87 to 1.15], Standard Error of Mean 0.072

8. Secondary Outcome: Proportion of Patients Dispensed an OAC Within One Year
Description: Evaluate the impact of the patient and provider education interventions on time to first OAC dispensing (prescription fill)
Time Frame: Outcome assessed at one year of follow-up time.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 23,546 | 23,787
Percent of participants | 9.84 [9.46 to 10.22] | 9.74 [9.36 to 10.12]
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.808, fixed-effect meta-analysis; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.95 to 1.07], Standard Error of Mean 0.029

9. Secondary Outcome: Number of Days Covered by OAC Dispensing
Description: Evaluate the impact of the patient and provider education interventions on proportion of days covered by OAC dispensings (prescription fills)
Time Frame: Outcome assessed at one year of follow-up time.
Population: Number of days on an OAC during all follow-up time among those initiated on OAC
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 2,678 | 2,673
days | 166.48 (129.75) | 168.15 (130.12)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.853, fixed-effect meta-analysis; Standardized Mean Difference (%) = -0.51, Standard Error of Mean 0.027

10. Secondary Outcome: Proportion of Patients on Oral Anticoagulation
Description: Evaluate the impact of the patient and provider education interventions on proportion of patients on oral anticoagulation at 12 months of follow-up
Time Frame: Outcome assessed at one year of follow-up time.
Population: Patients actively on an oral anticoagulant (OAC) at the end of follow-up among those treated for at least 1 day.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 2,074 | 2,095
Participants | 1,135 | 1,183
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.303, fixed-effect meta-analysis; Odds Ratio (OR) = 0.93, 95% CI 2-sided [0.82 to 1.06], Standard Error of Mean 0.066

11. Secondary Outcome: All-cause In-hospital Mortality Rates
Description: Evaluate the impact of the patient and provider education interventions on all-cause in-hospital mortality rates
Time Frame: Outcome assessed at one year of follow-up time.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention | Control
Number analyzed (Participants) | 22,964 | 23,232
Participants | 492 | 482
Statistical Analysis 1: Comparison: Intervention vs Control; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.649, fixed-effect meta-analysis; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.91 to 1.16], Standard Error of Mean 0.063

12. Secondary Outcome: Health Care Utilization for AF Patients
Description: Evaluate the impact of the patient and provider education interventions on health care utilization for AF patients, which would be reported as counts of number of health care utilization events (outpatient visits, days hospitalized, number of emergency department visits, etc.)
Time Frame: Outcome assessed at one year of follow-up time.
Measure: Mean (Standard Deviation); unit: Health care utilization events
Arm/Group | Intervention | Control
Number analyzed (Participants) | 23,546 | 23,787
Health care utilization events
  Total number of encounters at patient level | 40.40 (39.45) | 40.51 (39.51)
  Number of outpatient/ambulatory encounters | 38.17 (36.74) | 38.27 (36.81)
  Number of emergency department (ED) encounters | 0.66 (1.50) | 0.69 (1.75)
  Number of hospital admissions | 0.43 (0.91) | 0.44 (0.96)
  Number of institutional stays | 1.14 (3.36) | 1.10 (3.23)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.587, fixed-effect meta-analysis; Standardized Mean Difference (%) = -0.4998, Standard Error of Mean 0.009
Statistical Analysis 2: Comparison: Intervention vs Control; Test type: Superiority; p = 0.613, fixed-effect meta-analysis; Standardized Mean Difference (%) = -0.4655, Standard Error of Mean 0.009
Statistical Analysis 3: Comparison: Intervention vs Control; Test type: Superiority; p = 0.515, fixed-effect meta-analysis; Standardized Mean Difference (%) = 0.598, Standard Error of Mean 0.009
Statistical Analysis 4: Comparison: Intervention vs Control; Test type: Superiority; p = 0.018, fixed-effect meta-analysis; Standardized Mean Difference (%) = -2.17, Standard Error of Mean 0.009
Statistical Analysis 5: Comparison: Intervention vs Control; Test type: Superiority; p = 0.956, fixed-effect meta-analysis; Standardized Mean Difference (%) = 0.050, Standard Error of Mean 0.009

13. Secondary Outcome: Health Care Utilization for AF Patients, Days
Description: as for outcome 12
Time Frame: Outcome assessed at one year of follow-up time.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Intervention | Control
Number analyzed (Participants) | 23,546 | 23,787
days
  Days from modified intention-to-treat (mITT) start date to first outpatient/ambulatory encounter | 32.36 (47.99) | 32.76 (49.42)
  Number of days hospitalized | 3.01 (9.74) | 3.10 (9.27)
Statistical Analysis 1: Comparison: Intervention vs Control; Test type: Superiority; p = 0.279, fixed-effect meta-analysis; Standardized Mean Difference (%) = -1.018, Standard Error of Mean 0.009
Statistical Analysis 2: Comparison: Intervention vs Control; Test type: Superiority; p = 0.143, fixed-effect meta-analysis; Standardized Mean Difference (%) = -1.347, Standard Error of Mean 0.009

ADVERSE EVENTS:
Time Frame: Adverse events listed as secondary outcome measures in the protocol were assessed at 12 months following baseline. Adverse events were also passively monitored using a free telephone hotline, for 31 months following baseline for each participant
Description: We did not actively collect information about adverse events other than those listed as secondary outcome measures in the protocol. There were one or two sites that had no adverse events or just one event in either or both arms, so there was no estimated effect size/variance from the multivariable models at the site level. Depending on the specific outcome, either one or two sites did not contribute to the fixed-effect meta-analysis as there was no estimated effect size or variance to include.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 493/23546 | 483/23787
Serious Adverse Events (participants affected / at risk) | 737/23546 | 760/23787
Other Adverse Events (participants affected / at risk) | 0/23546 | 0/23787
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intervention (N=23546) | Control (N=23787)
Hospitalization for ischemic stroke or unknown stroke (Vascular disorders) | 343 | 375
Hospitalization for hemorrhagic stroke (Vascular disorders) | 82 | 65
Hospitalization for ischemic or hemorrhagic stroke (Vascular disorders) | 422 | 436
Hospitalization for ischemic or hemorrhagic stroke or systemic embolism (Vascular disorders) | 444 | 453
Hospitalization for ischemic or hemorrhagic stroke or systemic embolism or bleeding (Vascular disorders) | 737 | 760
Hospitalization for Bleeding (Vascular disorders) | 384 | 386

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-07): https://cdn.clinicaltrials.gov/large-docs/73/NCT03259373/Prot_001.pdf
  • Statistical Analysis Plan (2020-04-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT03259373/SAP_000.pdf